CLINICAL TRIAL: NCT05775146
Title: Phase II Single Arm Feasibility Trial to Evaluate Stereotactic Ablative Radiation of Metastases for the Management of Colorectal Cancer With Synchronous Oligo-metastases in Liver
Brief Title: SBRT of Metastases Following Neo-adjuvant Treatment for Colorectal Cancer With Synchronous Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0023
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Liver Metastasis Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT to the metastatic liver +/- lung lesions (Experimental): All rectal cancer patients included in the trial will receive short course radiation to the pelvis (with 25 Gy in 5 fractions) followed by chemotherapy with either 6 cycles of 3 weekly CAPOX chemotherapy or 9 cycles of 2 weekly FOLFOX. All colon cancer patients will receive 6 cycles of 3 weekly CAPOX or 9 cycles of 2 weekly FOLFOX. Patients will proceed for SBRT to the metastatic liver +/_ lung lesions and resection of the colorectal primary. Treatment planning is to be done using CT simulation or conventional simulation (Fluorocscopy) as per institutional practice. Simple beam arrangements, such as parallel opposed beams, are favored wherever possible.
  Interventions: Radiation: stereotactic body radiation treatment (SBRT)

INTERVENTIONS:
Radiation: stereotactic body radiation treatment (SBRT) — SBRT uses 3D imaging to target high doses of radiation to the affected area. There is very little damage to the surrounding healthy tissue. SBRT works by damaging the DNA of the targeted cells. Then, the affected cells can't reproduce, which causes tumors to shrink.

SUMMARY:
The purpose of this study is to prospectively evaluate the feasibility of SBRT for the management of synchronous oligo metastatic liver metastases from colorectal cancers.

DETAILED DESCRIPTION:
This will be a phase II feasibility trial to evaluate ablative radiation for the management of colorectal cancer with potentially resectable/ablatabale synchronous oligo-metastases.

In this study, following completion of the neo-adjuvant component of treatment, patients will be re-staged (as is the current standard of care) and can then proceed for SBRT to the liver lesion. Patients who may have responded very well to the systemic treatment with no-residual disease on re-staging imaging, will use pre-treatment imaging for target delineation. The advantage of SBRT is in the minimally invasive approach to treatment that may be associated with lower morbidity, better quality of life and post treatment morbidity, as well as being significantly less expensive.

The planned course of the neo-adjuvant component of treatment for this study will reflect the NCCN (National Comprehensive Cancer Network) guidelines and will treat rectal cancer patients with a short course of radiation followed by 6-9 cycles of a combination chemotherapy regimen.

For the colon cancer group of patients, all patients will receive 6-9 cycles (2-3 months) of neo-adjuvant systemic chemotherapy as per current standard of care.

Patients with non-progressive disease at that point, will have SBRT for the metastatic lesion followed by surgery for the primary rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG (Eastern Cooperative Oncology Group) 0-2
* Able to provide written informed consent
* 1-5 Liver lesions with max size of ≤5cm for a single lesion and restricted to one lobe of liver; deemed at Multi-Disciplinary Tumor Board (MDT) to be potentially amenable for SBRT with curative intent
* Liver lesion identified within 3 months of diagnosis of primary and deemed at Multi-Disciplinary Tumor Board (MDT) to be potentially amenable for SBRT with curative intent
* Plan for resection of primary with curative intent
* Patients with liver metastases and potentially resectable/ablatable lung mets can be included.
* Colon cancer patients who have undergone upfront resection of primary colonic lesion can be included
* Able and willing to comply with the terms of the protocol including health-related quality of life (HRQoL) questionnaires
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
* Females must not be breastfeeding
* Male patients should agree to not donate sperm during the study

Exclusion Criteria:

* Extra-hepatic metastases (except potentially resectable lung mets)
* Not a suitable candidate for liver resection surgery
* Not a suitable candidate for SBRT
* Past history of cancer within 5 years (except basal cell carcinoma)
* Patients who have undergone previous surgery or ablation for liver lesions
* Planned simultaneous resection of primary and liver metastases
* Pregnancy
* Patients with Child-Pugh C and documented cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of diagnosis upto 24 months in follow up
  Defined as Time from diagnosis to disease progression at any site or death

SECONDARY OUTCOMES:
Quality of Life (QOL)C309v3 | Baseline QOL will be assessed upto 24 months follow up
  To study the Quality of Life as measured by QLQ (quality of life questionnaire)-C309v3)
Quality of Life (QOL)EORTC | Baseline QOL will be assessed upto 24 months follow up
  To study the Quality of Life as measured by QLQ (quality of life questionnaire)- EORTC CR29 Questionnaire
Cancer Specific Survival (CSS) | Upto 24 months
  Defined as the time from diagnosis to death due to the cancer
Overall Suvival(OS) | Expected to be within 3 months post treatment
  Defined as the time from diagnosis to death due to any cause .
Toxicity Assessment | Toxicity assessment will be done upto 24 months in follow up
  Treatment related toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5

OTHER OUTCOMES:
Exploratory endpoints/outcomes. To identify blood biomarkers that can correlate with disease events | Blood samples will be collected at baseline upto 24 months in follow up
  Blood samples will be compared between the baseline and subsequent samples for changes in the expression levels of specific markers that may be associated with metastases and treatment response. These include circulating cell free DNA and exosomes. Carcino Embryonic Antigen (CEA) levels in blood will also be analysed. Micro Satellite Instability (MSI) pattern in the tumor tissue will be evaluated in the pathological tissue

CONTACTS AND LOCATIONS:
Overall Officials: Aswin Abraham, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No